CLINICAL TRIAL: NCT05772559
Title: Acute Myeloid Leukemia At Initial Diagnosis and/or Relapse in Children, Teenagers and Young Adults: Molecular Profiling, Multidrug Testing and MSC Interaction Studies - ALARM3
Brief Title: Acute Myeloid Leukemia At Initial Diagnosis and/or Relapse in Children, Teenagers and Young Adults: Molecular Profiling, Multidrug Testing and MSC Interaction Studies
Acronym: ALARM3
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP220571
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Acute Myeloid Leukemia; Genetic Predisposition to Disease
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1 : Patients with acute myeloid leukemia: Patients with acute myeloid leukemia at initial diagnosis or relapse, aged less than 25 years
  Interventions: Other: Collection of blood sample of bone marrow (cohort 1)
- Cohort 2 : Patients with genetic predisposition to develop acute myeloid leukemia
  Interventions: Other: Collection of blood sample of bone marrow (cohort 2 and 3)
- Cohort 3 : Patients who undergo bone marrow aspirate: Patients who undergo bone marrow aspirate as part of standard of care but without AML nor predisposition to develop AML, as controls
  Interventions: Other: Collection of blood sample of bone marrow (cohort 2 and 3)

INTERVENTIONS:
Other: Collection of blood sample of bone marrow (cohort 1) — * 3 additional tubes of blood sample (cohort 1), at diagnosis and upon relapse if relapse occurs
  * Bone marrow aspirate : 3 additional tubes (cohort 1), at diagnosis and upon relapse if relapse occurs
  Groups: Cohort 1 : Patients with acute myeloid leukemia
Other: Collection of blood sample of bone marrow (cohort 2 and 3) — * 1 additional tube of blood sample (cohort 2 and 3 at inclusion)
  * Bone marrow aspirate: 1 additional tube (cohort 2 and 3 at inclusion)
  Groups: Cohort 2 : Patients with genetic predisposition to develop acute myeloid leukemia; Cohort 3 : Patients who undergo bone marrow aspirate

SUMMARY:
Pediatric acute myeloid leukemias are disease with poor prognosis (overall survival of 60-75%) and high relapse rate of 35-45% require further understanding of the underlying biological mechanisms.

The main objective of this study is to establish a biological collection to evaluate the genomic profiling of leukemic cells from primary blasts at diagnosis and/or relapse to improve identification of the main genetic hits involved in resistance and could predict a high risk of relapse. Other objectives include the study of bone marrow mesenchymal stem cells and ex vivo drug testing.

ELIGIBILITY:
Inclusion Criteria:

* 0-25 years old
* Newly diagnosed de novo or secondary Acute Myeloid Leukemia (AML) or
* Relapsed or refractory AML or
* Patients with genetic predisposition to develop AML or
* Patients without haematological malignancy nor AML genetic predisposition syndrome who undergo bone marrow aspirate as part of standard of care
* Signed informed consent of parents for patients aged less than 18 years old or signed informed consent of the patient for patients aged 18 and over.

Exclusion Criteria:

* Refuse to participate
* Chronic myeloid leukemia (CML)
* Lack of health insurance (French social security)
* Under protection (tutelle, curatelle or sauvegarde de justice)
* Pregnancy or breastfeeding

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children or young adult with Newly diagnosed de novo or secondary Acute Myeloid Leukemia (AML) or Relapsed or refractory AML or patients with genetic predisposition to develop AML or patients without haematological malignancy nor AML genetic predisposition syndrome who undergo bone marrow aspirate as part of standard of care
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2033-05-31 (Estimated); Study Completion 2033-05-31 (Estimated)

PRIMARY OUTCOMES:
Number of somatic mutations in leukemic cells between diagnosis and relapse identified by Next-Generation Sequencing (NGS) | Up to 5 years

SECONDARY OUTCOMES:
Cumulative incidence of relapse (CIR) from remission status. | Up to 5 years
  Relapse is defined as:
  Bone marrow blasts ≥ 5% and/or evidence of extramedullary disease
Event Free Survival (EFS) | Up to 5 years
  Event Free Survival (EFS) is defined as the time from start of chemotherapy to failure, relapse, or death which ever occurs first
Disease Free Survival (DFS) | Up to 5 years
  Disease Free Survival (DFS) is defined as the time from remission status to relapse or death.
Number of mutations identified by WGS | Up to 5 years
  Number of mutations identified by Whole-Genome-Sequencing (WGS) as compared to Next-Generation Sequencing (NGS) in leukemic cells
Expression profile (transcriptome) of mesenchymal stem cells | Up to 5 years
  Expression profile (transcriptome) of mesenchymal stem cells at AML diagnosis and relapse compared to age matched controls without AML
Engraftment rate of primary leukemic cells | Up to 5 years
  Engraftment rate of primary leukemic cells in Patient-derived xenografts (PDX) or other experimental models
Matched rate of genetic mutational (or expression) profile between derived cells from experimental models to primary leukemic cells | Up to 5 years
Comparison of LSC signature profile of leukemic primary blasts at diagnosis and at relapse | Up to 5 years
Cumulative incidence of relapse according to LSC signature profile of leukemic primary blasts at diagnosis and at relapse | Up to 5 years
  Cumulative incidence of relapse according to Leukemic Stem Cell (LSC) signature profile of leukemic primary blasts at diagnosis and at relapse
EFS according to LSC signature profile of leukemic primary blasts at diagnosis and at relapse | Up to 5 years
  Event Free Survival according to Leukemic Stem Cell (LSC) signature profile of leukemic primary blasts at diagnosis and at relapse
DFS according to LSC signature profile of leukemic primary blasts at diagnosis and at relapse | Up to 5 years
  Disease-Free Survival (DFS) according to Leukemic Stem Cell (LSC) signature profile of leukemic primary blasts at diagnosis and at relapse
Ex vivo multidrug testing profile of leukemic primary blasts | Up ot 5 years
  Comparison of ex vivo multidrug testing profile of leukemic primary blasts at diagnosis and relapse
Cumulative incidence of relapse according to ex vivo multidrug testing profile of leukemic primary blasts at diagnosis and relapse | Up to 5 years
EFS according to ex vivo multidrug testing profile of leukemic primary blasts at diagnosis and relapse | Up to 5 years
  Event-Free Survival according to ex vivo multidrug testing profile of leukemic primary blasts at diagnosis and relapse
DFS according to ex vivo multidrug testing profile of leukemic primary blasts at diagnosis and relapse | Up to 5 years
  Disease Free Survival according to ex vivo multidrug testing profile of leukemic primary blasts at diagnosis and relapse
Mutational profile of patients | Up ot 5 years
  Comparison of mutational profile of patients with a predisposition syndrome compared to mutational profile of patients with AML at diagnosis and relapse
Percentage of MRD clearance | Up to 5 years
  MRD clearance is defined as MRD below 10-3 Evaluated by flow cytometry and high sensitivity NGS (defined as MRD below 10-4) after each chemotherapy course
Cumulative incidence of relapse according to MRD clearance | Up to 5 years
  Evaluated by flow cytometry at a sensitivity threshold of 10-3
EFS according to MRD clearance | Up to 5 years
  Evaluated by flow cytometry at a sensitivity threshold of 10-3
DFS according to MRD clearance | Up to 5 years
  Evaluated by flow cytometry at a sensitivity threshold of 10-3
Cumulative incidence of relapse according to MRD clearance | Up to 5 years
  Evaluated by high sensitivity NGS at a threshold of 10-4
EFS according to MRD clearance | Up to 5 years
  Evaluated by high sensitivity NGS at a threshold of 10-4
DFS according to MRD clearance | Up to 5 years
  Evaluated by high sensitivity NGS at a threshold of 10-4

CONTACTS AND LOCATIONS:
Locations (28):
- France (28):
  - CHU Amiens Picardie site Sud, Amiens
  - CHU Angers, Angers
  - Hopital Minjoz, Besançon
  - CHU Pellegrin, Bordeaux
  - CHRU Morvan, Brest
  - CHU Caen, Caen
  - CHU Estaing, Clermont-Ferrand
  - CHU Francois Mitterand, Dijon
  - CHU Grenoble, Grenoble
  - CHU de la Réunion, La Réunion
  - Hopital Jeanne de Flandre - CHRU, Lille
  - CHU Limoges, Limoges
  - HCL Lyon, Lyon
  - Hôpital d'Enfants de la Timone, Marseille
  - CHU Montpellier, Montpellier
  - CHRU Nancy- Hopitaux de Brabois, Nancy
  - CHU Nantes, Nantes
  - CHU Nice, Nice
  - Hopital Robert Debré, Paris
  - Hopital Trousseau, Paris
  - CHU Poitiers, Poitiers
  - Hopital Américain, Reims
  - CHU Hopital Sud, Rennes
  - CHU Rouen, Rouen
  - CHU Saint Etienne, Saint-Etienne
  - Hopital Hautepierre, Strasbourg
  - CHU Toulouse, Toulouse
  - CHRU Tours, Tours